CLINICAL TRIAL: NCT00095407
Title: The Functional Anatomy of Personality Trait Knowledge: an fMRI Study
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050018; 05-N-0018
Record Dates: First submitted 2004-11-03; First posted 2004-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-12-29

CONDITIONS: Healthy
Keywords: Social Cognition; Semantic Memory; Prefrontal Cortex; Temporal Cortex; Conceptual Self

SUMMARY:
This study will identify the regions of the brain that are involved in personality trait knowledge-that is, what a person knows about aspects of personality such as "generous," "honest," and others. It will also examine brain areas relating to a person's knowledge of how likeable those personality traits are, being familiar with the traits, and the degree of associating such traits with one's self. There has not been any previous study, through modern imaging techniques, on the location of the brain and the concepts of personality traits.

Patients ages 21 to 65 who are in good health, are right handed, and native speakers of English may be eligible for this study. Pregnant women are not eligible. There will be 200 participants involved in pencil-and-paper or computer tasks. Also, there will be three functional magnetic resonance imaging (fMRI) experiments with 32 participants. Patients may participate in up to three fMRI experiments.

Patients will be recruited through NIH's Normal Control Database. They would need to have had a neuroexamination conducted by an NIH doctor within the last year. Patients will be interviewed for any medical, neurological, or psychological condition that would make it difficult to read the fMRI results. Depending on the studies that patients take part in, they will have different questionnaires to complete. They may also perform a computerized test that measures word associations. These tests will take about 1 to 2 hours.

The technique of MRI uses a strong magnetic field and radio waves to obtain images of body organs and tissues. During the initial MRI scan, patients will lie still on a table that will slide into the enclosed tunnel of the scanner. They will be in the scanner not longer than 2 hours. During the procedure, they may be asked to lie as still as possible for up to 1 hour at a time. As the scanner takes pictures, patients will hear knocking or beeping sounds, and they will wear earplugs to reduce the noise. Patients will be able to communicate with the MRI staff at all times during the scan, and they may ask to be moved out of the machine at any time. Then the functional MRI (fMRI) scan will involve taking pictures of the brain while patients are performing tasks. All the tasks will be explained, and patients will have the chance to practice them before entering the scanner. For this activity, patients will be asked to make decisions about what they are seeing in the tasks presented to them. They will decide "yes" and "no" by pressing a left or right button. This scan will take about 1 hour. Afterward, patients may be asked to fill out written questionnaires or to perform reaction time tasks by using a computer.

This study will not have a direct benefit for participants. However, it is hoped that information gained will enhance researchers' understanding about which areas of the brain are necessary to perform certain tasks.

DETAILED DESCRIPTION:
Objective. The purpose of the protocol is to identify the brain regions involved in personality trait knowledge, associated affective valence and person-trait associations. We propose using parametric event-related fMRI in addition to classical reaction time measures, to answer the question of whether a specialized neural system is involved in semantic processing of personality trait concepts. We will apply methods that have been used in previous investigations to identify category-specific semantic (meaning) systems for living and non-living objects.

Study Population. Healthy, normal adult, right-handed volunteers will be studied during functional neuroimaging and in behavioral pre-tests.

Design. Behavioral pre-tests (N=200 subjects) are used to obtain psycholinguistic stimulus parameters used in the fMRI experiments. Three parametric event-related functional MRI experiments (for a total of 104 subjects) using personality trait concept words as main input stimuli will be conducted.

Outcome Measures. The data collected will consist of questionnaire results, behavioral measures of cognitive performance and corresponding fMRI images. The results gained from this protocol will be of value in advancing the neuroscience of person perception and social cognition.

ELIGIBILITY:
* INCLUSION CRITERIA:

In all the studies, subjects will consist of healthy, native English-speaking, right-handed volunteers, as measured by the Edinburgh Handedness Inventory (Oldfield, 1971). Subjects will range in age from 21 to 65 years old and they will be included regardless of race and gender.

EXCLUSION CRITERIA:

Non-native English speakers and non-right handers will be excluded as mentioned above, as will non-neurologically normal volunteers. Subjects younger than 21 and older than 65 will be excluded. A urine pregnancy test will be employed with all women of childbearing age no more than 24 hours prior to the MRI. The results must be negative in order to proceed with the MRI.

Participants with any of the following: aneurysm clip; implanted neural stimulator; implanted cardiac pacemaker or auto-defibrillator; cochlear implant; ocular foreign body, e.g. metal shavings; permanent eyeliner; insulin pump; or irremovable body piercing will be excluded from the study due to the possible dangerous effects of the magnet upon metal objects in the body. Participants taking central nervous system active medications will be excluded.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2004-10-29; Study Completion 2011-12-29

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Adolphs R. Cognitive neuroscience of human social behaviour. Nat Rev Neurosci. 2003 Mar;4(3):165-78. doi: 10.1038/nrn1056. PMID 12612630
- [Background] Altshuler LL, Bartzokis G, Grieder T, Curran J, Mintz J. Amygdala enlargement in bipolar disorder and hippocampal reduction in schizophrenia: an MRI study demonstrating neuroanatomic specificity. Arch Gen Psychiatry. 1998 Jul;55(7):663-4. doi: 10.1001/archpsyc.55.7.663. No abstract available. PMID 9672058
- [Background] Ashburner J, Friston KJ. Voxel-based morphometry--the methods. Neuroimage. 2000 Jun;11(6 Pt 1):805-21. doi: 10.1006/nimg.2000.0582. PMID 10860804